CLINICAL TRIAL: NCT06875570
Title: Effects of a 12-Week Combined Training Protocols on Aerobic Fitness, Technical Skills, and Psychophysiological Responses in Young Recreational Volleyball Players
Brief Title: Effects of Combined Training Protocol in Volleyball Players
Acronym: SSGs+PL+JR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Neslihan AKÇAY, Assoc. Prof. Dr., Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKarabuk-4
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Volleyball; Performance; Training; Technical Skills
Keywords: Volleyball; Small Sided Games; Pliometric; Jump rope

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were strictly separated and think their intervention is the main intervention. The same is true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pliometric Training (Experimental): Players will receive a Plyometric training program at the beginning of the Volleyball training session for a period of 15 minutes, two days a week.
  Interventions: Other: Pliometric Training
- Jump Rope training (Experimental): Players will receive a jump rope training program at the beginning of the volleyball training session for 15 minutes, two days a week.
  Interventions: Other: Jump Rope Training
- Small Sided Games (Experimental): More complex, skill-based conditioning exercises for volleyball are small-sided games (2v2, 3v3) and competition drills (6v6).
  Interventions: Other: Small Sided Games

INTERVENTIONS:
Other: Pliometric Training — The full intervention program will cover 12 weeks in the season. Prior to training, players will be instructed to warm-up for ten minutes with general running exercises and dynamic stretching. The plyometric training intervention will consist of 5 exercises performed in the following order: Leap forward and backward on the line, leap sideways on the line, double leg knee to chest, split squat jump, and squat jump (Bavli, 2012). A volleyball coach will monitor the whole training.
  Arms: Pliometric Training
Other: Jump Rope Training — The entire intervention program will last for 12 weeks during the season. Before training, players will be instructed to warm up with general running exercises and dynamic stretching for ten minutes. The jump rope intervention will consist of 5 exercises performed in the following order: basic jump step, double leg double jump, double leg jump left and right, double leg jump forward and backward, and scissor steps (Trecroci et al., 2015). Each exercise will be performed by all participants using a jump rope with the same characteristics in terms of weight (e.g. 230g), length (e.g. shoulder size) and material (e.g. PVC, Polyvinyl Chloride). A metronome speed of 120 beats per minute will be used to ensure equal exercise intensity in both exercise programs Furthermore, a volleyball coach will monitor the entire workout.
  Arms: Jump Rope training
Other: Small Sided Games — More complex, skill-based conditioning exercises for volleyball are small-sided games (2v2, 3v3) and competition drills (6v6). Although the duration of each rally in these drills is not controlled by the coach, the total duration of the drill will be recorded to aid in-session and inter-session planning. Total repetitions will be easily measured by adding up the total points played in the rally and then multiplying by the number of rallies per point. The coach will create an emotionally intense environment by applying a scoring system (e.g. team winning 2 out of 3 rallies gets 1 big point, 5 seconds rest) and encouraging the players (Trajkovic et al., 2012).
  Arms: Small Sided Games

SUMMARY:
The 12-week training will take place during the preparation period. At the beginning and end of the 12-week period, vertical jump test, 60 seconds countermovement jump (CMJ) test, change of direction (T-Agility) test, sprint test, YO-YO (level-1) test will be applied in terms of performance test. In terms of skill testing, service test and spiking test protocols will be applied. Players will perform plyometric (PL) or jump rope (JR) training with the same amount of total training time in each training session. Rating of perceived exertion (RPE) will be obtained using (CR6-20). All players will also complete the short form of the physical activity enjoyment scale (PACES).

DETAILED DESCRIPTION:
There will be 12 weeks of training during the preparation period. Each daily training will start with a 10-minute standard warm-up consisting of running, dynamic stretching and sprinting with volleyball-specific technical movements integrated. After warm-up and Small Sided Games (2v2, 3v3, 4v4, 5v5), players will perform plyometric (PL) or jump rope (JR) training with the same amount of total training time in each training session. At the start of the 12-week period, the vertical jump and 60 second countermovement jump (CMJ) using a portable force plate (Smart Jump; Fusion Sport, Queensland, Australia), T-Agility change of direction and Sprint tests with timing gates (Smart Speed; Fusion Equipment, Brisbane, Australia) and Yo-Yo Intermittent Recovery Test Level 1 will be used for VO2max levels. Serve and Spiking Technical Skill Tests will be applied together with these. To minimise the negative effects of fatigue on psychological, physiological and performance responses, each training intervention will be performed at least 2 days apart. Rating of perceived exertion (RPE) will be obtained using the category ratio scale (CR6-20) to calculate the internal training load (ITL) immediately after the completion of each session. The scale will be introduced at baseline to familiarise players. All players will also complete the short form of the physical activity enjoyment scale (PACES). The scale consists of 8 items scored on a 1-7 Likert scale and has been validated as an indicator of Turkish youth's level of enjoyment of activity.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male volleyball athletes
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Being under 18 years old
* Having a chronic disease
* Contraindications for exercise

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump | From baseline assessment to 12 week follow-up assessment]
  Change in vertical jump (cm) is expected from baseline assessment to 12-week follow-up assessment
60s Countermovement Jump | From baseline assessment to 12 week follow-up assessment
  Change in countermovement jump (watts/kg) is expected from the baseline assessment to the 12-week follow-up assessment..
Change of Direction | From baseline assessment to 12 week follow-up assessment]
  Changes in change of direction times (sec) are expected from the baseline assessment to the 12-week follow-up assessment.
Sprint | From baseline assessment to 12 week follow-up assessment
  Change in Sprint (km/h) is expected from the baseline assessment to the 12-week follow-up assessment.
Yo-Yo Intermittent Recovery Test Level 1 | From baseline assessment to 12 week follow-up assessment
  A change in VO2max values from the baseline assessment to the 12-week follow-up assessment is expected.
Service | From baseline assessment to 12 week follow-up assessment
  A change in service test values from the baseline assessment to the 12-week follow-up assessment is expected.
Spiking | From baseline assessment to 12 week follow-up assessment
  A change in spiking test values is expected from the baseline assessment to the 12-week follow-up assessment.
Rating of Perceived Exertion (RPE) | From baseline assessment to 12 week follow-up assessment
  Changes in Rating of Perceived Exertion (RPE) are expected from the baseline assessment to the 12-week follow-up assessment. The scale has a range of 6-20 (CR20). Athletes will indicate whether they do not find exercise difficult (6) or find it difficult (20).
PAGES | From baseline assessment to 12 week follow-up assessment
  Changes are expected in the Enjoyment of physical activity scale (PACES) from the baseline assessment to the 12-week follow-up assessment. The scale consists of 8 questions with a score range of 1-7. Athletes will indicate whether they do not enjoy exercise (1) or enjoy it (7).

OTHER OUTCOMES:
Anthropometric Measurements 1 | Baseline
  Participants' height (cm) will assess by using a stadiometer (Holtain Stadiometer, England).
Anthropometric Measurements 2 | Baseline
  Body weight (kg) will asses by Inbody 270 (Biospace, California, USA)
Anthropometric Measurements 3 | Baseline
  Body mass index (BMI) (kg/m2) will asses by Inbody 270 (Biospace, California, USA).
Anthropometric Measurements 4 | Baseline
  Body fat percentage (%) will asses by Inbody 270 (Biospace, California, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Akçay, Doctorate, Study Chair — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fathi A, Hammami R, Moran J, Borji R, Sahli S, Rebai H. Effect of a 16-Week Combined Strength and Plyometric Training Program Followed by a Detraining Period on Athletic Performance in Pubertal Volleyball Players. J Strength Cond Res. 2019 Aug;33(8):2117-2127. doi: 10.1519/JSC.0000000000002461. PMID 29401199
- [Background] Ozer D, Duzgun I, Baltaci G, Karacan S, Colakoglu F. The effects of rope or weighted rope jump training on strength, coordination and proprioception in adolescent female volleyball players. J Sports Med Phys Fitness. 2011 Jun;51(2):211-9. PMID 21681154
- [Background] Voelzke M, Stutzig N, Thorhauer HA, Granacher U. Promoting lower extremity strength in elite volleyball players: effects of two combined training methods. J Sci Med Sport. 2012 Sep;15(5):457-62. doi: 10.1016/j.jsams.2012.02.004. Epub 2012 Apr 6. PMID 22484082